CLINICAL TRIAL: NCT01373528
Title: Impact of Topical Sinonasal Budesonide Irrigation on Hypothalamic-Pituitary-Adrenal (HPA) Axis Function
Brief Title: Impact of Topical Sinonasal Budesonide Irrigation on Hypothalamic-Pituitary-Adrenal Axis Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010249-01H
Record Dates: First submitted 2011-06-12; First posted 2011-06-15 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Rhinosinusitis
Keywords: Sinonasal Budesonide; Endoscopic sinus surgery; Hypothalamic-Pituitary-Adrenal Axis Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Budesonide (Experimental)
  Interventions: Drug: Budesonide irrigation

INTERVENTIONS:
Drug: Budesonide irrigation — A budesonide (1 mg) in saline (240 mL) irrigation solution is applied to the sinonasal cavities twice daily. 120 mL of the solution is applied via irrigation in the AM, and 120 mL again in the PM.

SUMMARY:
Chronic rhinosinusitis (CRS) is a complex inflammatory disease that is treated primarily with sinus surgery and the long-term use of topical steroid therapy. Budesonide irrigation is a common method of topical steroid treatment for these patients. However, the effects of budesonide irrigation on the hypothalamic-pituitary-adrenal (HPA) axis in patients with CRS following sinus surgery, is as of yet not defined. The objective of this study is to determine if topical sinonasal budesonide steroid irrigation leads to acute recoverable and/or long-term suppression of the HPA axis. Participants in this prospective cohort study will have CRS and have recently undergone endoscopic sinus surgery. They will also have had planned use of budesonide irrigations as their postoperative medical treatment. The acute effects of this treatment on the HPA axis will be evaluated using serial serum cortisol measurements both the day before and the day of the first budesonide irrigation. The long-term effect of sinonasal budesonide irrigation will be evaluated using both a pre- and post-treatment adrenocorticotropic hormone (ACTH) stimulation test as well as repeated urine free cortisol levels over the length of the study. The results will determine the need for additional steroids when patients stop treatment or with a physiologic stressful event.

DETAILED DESCRIPTION:
CRS is an inflammatory disease of the paranasal sinuses that is difficult to treat. Current treatment strategies rely upon medical treatment with the long-term daily use of a topical corticosteroid as its foundation. Once medical therapy becomes ineffective at controlling CRS and its resultant symptoms, surgical treatment is offered. Following surgery, patients must again continue with medical treatment to control the inflammation present in CRS. Previously, topical steroids could be applied using only a commercially prepared applicator that is effective at treating no more than the front of the nose and parts of the paranasal sinuses. However, relatively new nasal saline irrigation devices have made it possible to treat all of the paranasal sinuses. Corticosteroid medication can be added directly to the saline irrigation. In an operated patient the sinus openings have been greatly enlarged which then allows the irrigation to more effectively reach all of the paranasal sinuses. Therefore, irrigation with a corticosteroid solution allows for better delivery of the corticosteroid medication to treat the mucosal inflammation that is widely present. More effective treatment of the paranasal sinus inflammation thereby leads to improved control of inflammation and to the alleviation of patient symptoms such as chronic facial and dental pain, headache, obstructed nasal breathing, loss of smell and discharge from the nose. As of yet, with this method of treatment it has not been determined whether there is significant systemic absorption and a resultant suppression of the HPA axis.

The investigators hypothesize that:

1. a single 0.5 mg dose of budesonide will result in acute but recoverable suppression of pituitary adrenocorticotrophic hormone (ACTH) secretion with a resultant transient decrease in adrenal cortisol production; and that
2. the long term use of budesonide, 0.5 mg twice daily (BID), will result in a gradual and cumulative suppression of the HPA axis to the extent that significant hypocortisolism will be present when budesonide irrigation is discontinued necessitating replacement glucocorticoid therapy.

Specific Aim of Project This study will determine if there is acute recoverable and long-term suppression of the HPA axis when budesonide irrigations are used in patients with CRS following endoscopic sinus surgery. This important information is currently not available in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult patients (age ≥18) who are diagnosed with CRS
* Patient already determined to need surgical treatment having failed medical management
* Patients planned to be treated with budesonide irrigations as postoperative maintenance therapy

Exclusion Criteria:

* Patients with pre-operative symptoms and signs of HPA dysfunction
* Patients with signs and symptoms of untreated endocrine disorders such as hypothyroidism, hypopituitarism, hypogonadism. Screening for thyroid disease will be done with a TSH, T3 and free T4 for each participant.
* Patients with known history of liver disease or abnormal AST/ALT lab tests
* Any history of oral glucocorticoid use in the past 4 months
* Patients with a known history of glaucoma
* Patients with known tuberculosis (TB)- active or latent
* Patients taking drugs that affect cortisol synthesis (mifepristomine, itraconazole, ketoconazole, erythromycin, clarithromycin, cimetidine) or protein binding drugs (estrogens and androgens)
* A known sensitivity to topical budesonide
* Pregnant and/or breast feeding woman
* Presence of multiple co-morbidities such as poorly controlled diabetes, chronic renal failure, hepatic failure
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Serum cortisol levels before and after treatment | 12 months
ACTH stimulation test cortisol level | 12 months
Urinary Free Cortisol Levels | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kilty Shaun, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital Riverside Campus, Ottawa, Ontario, Canada